CLINICAL TRIAL: NCT06230510
Title: Milk Type in Toddlers (Milk-TOT) Study: Impact of Whole Versus Low-fat Milk on Child Adiposity, Health and Development
Brief Title: Milk-Tot Study: Impact of Whole Versus Low-fat Milk on Child Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Stanford University (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1757040; R01DK131217 (NIH)
Record Dates: First submitted 2023-12-11; First posted 2024-01-30 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two groups in parallel for one year.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole Milk (Experimental): Whole Milk consumption for one year
  Interventions: Behavioral: Introduction of Milk Type; Behavioral: Child Nutrition Counseling
- 1% Milk (Experimental): 1% Milk consumption for one year
  Interventions: Behavioral: Introduction of Milk Type; Behavioral: Child Nutrition Counseling

INTERVENTIONS:
Behavioral: Introduction of Milk Type — Beginning at approximately age 2, milk (equivalent to 2 cups/day) will be provided at no cost to the family for one year.
Behavioral: Child Nutrition Counseling — Parent/caregivers will receive quarterly phone-based counseling by a Registered Dietitian (RD) on how to introduce the toddler to the assigned milk and the importance of continuing to drink the assigned milk for the one year.

SUMMARY:
In the U.S. it is recommended that children consume whole cow's milk (3.5% fat) from ages 1 to 2 years to support rapid early growth and brain development, and then at age 2 years transition to low-fat (1%) or non-fat milk to reduce saturated fat and calorie intake. To date, few studies have examined the optimal milk type for children to prevent obesity. This randomized controlled trial will evaluate the effect of consumption of whole versus 1% milk on child adiposity.

DETAILED DESCRIPTION:
The prevalence of child obesity in the U.S. has tripled since the 1970s and excess weight gain - even in young children - is a precursor to adult obesity and associated co-morbidities. In the U.S. it is recommended that children consume whole cow's milk (3.5% fat) from ages 1 to 2 years to support rapid early growth and brain development, and then at age 2 years transition to low-fat (1%) or non-fat milk to reduce saturated fat and calorie intake. However, surprisingly few rigorous trials to support recommendations on optimal milk type have been conducted and existing observational studies paradoxically suggest that lower fat milk consumption is associated with increased adiposity in children. The effects of the types of fat found in milk on cardiometabolic disease risk have also been questioned. This randomized controlled trial will evaluate the effect of consumption of whole versus 1% milk on child adiposity and other health and developmental outcomes beginning after toddlers have successfully transitioned from breastmilk and/or formula to cow's milk at 2 years of age. Investigators will recruit 625 parents of toddlers and randomly assign 625 toddlers to either whole or 1% milk groups for 1 year (with estimated final sample size of 500). Our primary aim is to determine how milk fat type (whole versus 1%) consumed from age 2 to 3 years affects change in adiposity as measured by waist-to-height ratio (primary outcome), body mass index, tri-ponderal mass index, and waist circumference. Secondary aims are to evaluate how milk type consumed from age 2 to 3 years affects changes in milk, total and saturated fat, added sugars, and total energy intake and overall diet quality, as well as blood lipids and vitamin D status, and neurocognitive development. Results from the Milk-TOT Study can help pediatric health care providers give evidence-based dietary recommendations to improve child weight and health, and can inform the types of milk provided to participants in the federal nutrition programs which collectively provide milk to over half of all young children in the U.S.

ELIGIBILITY:
Inclusion Criteria:

Parents of children: 1) willing to be randomized to provide either only whole or 1% milk to their child for 1 year, 2) access to a smart phone and a tablet, laptop or computer with internet and email at home, 3) ability to speak and read English or Spanish for the purposes of receiving study communications and completing surveys and dietary assessments (to avoid needing to translate all study materials and have research staff fluent in other languages due to budget limits), 4) not planning to move outside of the San Francisco Bay Area or discontinue being child's primary caregiver for the next year (e.g., foster care, parent separation).

Exclusion Criteria:

Children: 1) <23 months or >48 months old at recruitment; 2) condition or medication that affects growth or daily feeding, or cardiometabolic health such as hypopituitarism, growth hormone deficiency, inborn error of metabolism, syndromic obesity, familial hypercholesterolemia, 3) weight-for-length or height below the 2nd percentile, 4) lactose intolerance, milk allergy or other dietary restrictions (e.g., vegan) that impact ability to consume dairy or otherwise limit dietary intake, 5) resides in more than one household (e.g., shared care by separated parents), 6) current participation in the Special Supplemental Nutrition Program for Women, Infants, and Children (WIC) (which provides milk as part of benefits), 7) not covered by public or private medical insurance (may reduce well-child doctor visits). If two eligible children are in a household, one will be randomly selected to participate.

Ages: 23 Months to 48 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 625 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in waist-to-height ratio | Baseline and 12-months after the start of the study.
  Waist-to-height ratios will be calculated using measured height in m and waist circumference in m.

SECONDARY OUTCOMES:
Change in body mass index z-score | Baseline and 12-months after the start of the study.
  BMI z-scores will be determined using measured height in m and weight in kg to calculate kg/m^2, and Centers for Disease Control and Prevention (CDC) growth curves.
Change in tri-ponderal mass index | Baseline and 12-months after the start of the study.
  Try-ponderal mass index (TMI) will be determined using measured height in m and weight in kg to calculate kg/m^3.
Change in waist circumference z-score | Baseline and 12-months after the start of the study.
  Waist circumference z-scores will be determined using measured waist circumference and CDC growth curves.
Change in dietary intake | Baseline and 12-months after the start of the study.
  Energy (kcals/day), milk (cups/day and %kcals), total dairy (cups/day and %kcals), total fat (g/day and %kcals), saturated fat (g/day and %kcals), added sugars (g/day and %kcals) and calcium (mg/day) intake will be measured using 24-hour recalls.
Change in diet quality | Baseline and 12-months after the start of the study.
  Diet quality will be measured using the healthy eating index-2020 from 24-hour recalls.
Change in blood measures | Baseline and 12-months after the start of the study.
  Lipid concentrations, glucoregulatory indices, and 25(OH)D concentrations will be measured in a morning blood draw.
Change in brain growth | Baseline and 12-months after the start of the study.
  Head circumference z-scores will be determined using measured head circumference in cm and CDC growth curves.
Change in neurocognitive development | Baseline and 12-months after the start of the study.
  Cognitive, communication and physical development scores will be determined using the Developmental Assessment of Young Children-2 tool.

CONTACTS AND LOCATIONS:
Overall Officials: Lorrene Ritchie, PhD, Principal Investigator — Nutrition Policy Institute
Locations (1):
- Nutrition Policy Institute, University of California Agriculture and Natural Resources, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: No